CLINICAL TRIAL: NCT01523743
Title: Quality of Life Intermittent Catheter Study - A Prospective, Randomized, Cross-over, Multicenter Study Comparing Quality of Life Using Compact Versus Standard Urinary Intermittent Catheters
Brief Title: Quality of Life Intermittent Catheter Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP220
Record Dates: First submitted 2012-01-09; First posted 2012-02-01 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Neurogenic Bladder Dysfunction Nos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compact catheter (Experimental): Compact intermittent catheter
  Interventions: Device: SpeediCath Compact
- Standard Care (Active Comparator): Standard Care: Coated intermittent catheter normally used by subject
  Interventions: Device: Standard care

INTERVENTIONS:
Device: SpeediCath Compact — The SpeediCath Compact intermittent catheter is used for single-use urinary bladder drainage through the urethra.
  Other Names: SpeediCath®Compact Male, for male participants; SpeediCath®Compact Female, for female participants
  Arms: Compact catheter
Device: Standard care — The coated intermittent catheter normally used by subject
  Arms: Standard Care

SUMMARY:
The purpose of this study is to compare compact intermittent catheters with standard coated intermittent catheters with regard to quality of life, using the Intermittent Self-Catheterisation Quality of life Measure.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age
* Has given written informed consent
* Has neurogenic bladder dysfunction
* Has used coated intermittent catheter as primarily bladder emptying method for at least 6 months
* Is able to self-catheterise
* Is able to use SpeediCath® compact catheters
* If spinal cord injury subject, injury must have occurred more than 12 months ago
* Covered by Social security system

Exclusion Criteria:

* Has used SpeediCath® compact catheters (not including screening for this investigation)
* Is admitted to rehabilitation centre
* Subjects using primarily catheter sets
* Is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Chartier-Kastler, Proff, Principal Investigator — Hôpital Raymond poincarè, Service d'Urologie, Garches, France
Locations (11):
- Denmark (3):
  - PrivatHospitalet Danmark, privat hospital,, Charlottenlund
  - Rigshospitalet, Urology clinic,, Copenhagen
  - CCBR Vejle, Clinical research site,, Vejle
- France (4):
  - Hôpital Tenon, Neuro-Urology and perineal explorations department,, Paris, Cedex 20
  - Hôpital Raymond Poincaré, Urology clinic, Garches
  - Hôpital Léon Berard, Rehabilitation clinic,, Hyères
  - Hôpital Henry Gabrielle, Urology clinic,, Saint-Genis-Laval
- University Heidelberg, Neuro-Urology clinic,, Heidelberg, Germany
- St. Olavs Hospital HF, Neurologi clinic,, Trondheim, Norway
- Sweden (2):
  - Gävle sjukhus, Urology clinic,, Gävle
  - Rehab Station Stockholm,, Stockholm

REFERENCES:
- [Derived] Prieto JA, Murphy CL, Stewart F, Fader M. Intermittent catheter techniques, strategies and designs for managing long-term bladder conditions. Cochrane Database Syst Rev. 2021 Oct 26;10(10):CD006008. doi: 10.1002/14651858.CD006008.pub5. PMID 34699062

RESULTS

PARTICIPANT FLOW:
Groups:
- First Compact Catheter, Then Standard Care: First period: Compact intermittent catheter from Coloplast. Second period: Standard Care: Coated intermittent catheter normally used by subject
- First Standard Care; Then Compact Catheter: First period: Standard Care: Coated intermittent catheter normally used by subject Second period: Compact catheter: Compact intermittent catheter from Coloplast
Period: Period 1
Arm/Group | First Compact Catheter, Then Standard Care | First Standard Care; Then Compact Catheter
Started | 63 | 62
Completed | 53 | 60
Not Completed | 10 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Felt unable to empty bladder | 1 | 0
Period: Period 2
Arm/Group | First Compact Catheter, Then Standard Care | First Standard Care; Then Compact Catheter
Started | 53 | 60
Completed | 52 | 58
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The ITT population consistsed of 118 subjects.
Groups:
- All Study Participants: 125 subjects were randomized in this study, however 7 subjects discontinued only providing baseline data and were therefore excluded from the ITT population as they did not contribute with any endpoint data.
  The baseline and analysis data are based on the ITT population.
Arm/Group | All Study Participants
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 103
Region of Enrollment [Number; unit: participants]
  France | 40
  Denmark | 27
  Norway | 5
  Germany | 18
  Sweden | 28

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life (0-100 Point)
Description: Difference in intermittent self-catheterisation quality of life measure, comparing compact versus standard urinary intermittent catheters The range of the scale is 0-100 where a high score indicating a high level of Quality of Life.
Time Frame: 6 weeks
Population: The primary analysis was based on the ITT population which included 118 subjects. 7 subjects were excluded from the ITT population. They were excluded because they discontniued the investigation and only baseline data was collected from them. Furthermore, not all subjects in the ITT population answered the QoL questionaire for both products.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Compact Catheter | Standard Care
Number analyzed (Participants) | 112 | 114
units on a scale | 76.8 (14.5) | 59.8 (19.3)

ADVERSE EVENTS:
Arm/Group | Compact Catheter | Standard Care
Serious Adverse Events (participants affected / at risk) | 3/123 | 2/115
Other Adverse Events (participants affected / at risk) | 16/123 | 14/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compact Catheter (N=123) | Standard Care (N=115)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neuropathic pain (Nervous system disorders) | 1 (1) | 0 (0)
Pleuritis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compact Catheter (N=123) | Standard Care (N=115)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
UTI (Infections and infestations) | 2 (2) | 5 (5)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cold (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Neuropathic pain (Nervous system disorders) | 0 (0) | 1 (1)
Anal hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Planned plastic surgery of ulcer (Surgical and medical procedures) | 0 (0) | 1 (1)
Urethral sensitivity when Catheter removed (Surgical and medical procedures) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Pain in hands (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abscess tooth and gingival (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Ischial pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tendinophaty (Nervous system disorders) | 0 (0) | 1 (1)
Skin herpes (Infections and infestations) | 1 (1) | 0 (0)
Spasticity of legs (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days